CLINICAL TRIAL: NCT04352426
Title: Effectiveness of Symptom-limited Stair-climbing Test in the Determination of the Exercise Capacity of Patients With Chronic Heart Failure
Brief Title: Symptom-limited Stair Climbing Test in Heart Failure
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Other Study IDs: busra.alkan
Record Dates: First submitted 2020-04-06; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; exercise capacity; symptom-limited stair-climbing test
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Exercise Test — Tests were conducted to evaluate exercise capacity.

SUMMARY:
Aims: To assess the efficacy of symptom-limited stair-climbing test (SLSCT), in determining the exercise capacities of patients with chronic heart failure (CHF) in comparison with cardiopulmonary exercise test (CPET) and 6-minute walk test(6MWT) and to interpret the results according to the clinical status of the patients.

Methods: Thirty-one patients, aged 50-75 years, with stage II-III CHF according to the New York Heart Association Classification and left ventricular ejection fraction (LVEF) of ≤45% were included. The demographic and clinical characteristics of the patients were recorded. Exercise capacity was assessed by SLSCT, 6MWT, and CPET. The duration of patients' performance in the test, reasons for ending the test and predicted maximal oxygen consumption (VO2max) were recorded. Heart rate (HR), blood pressure (BP), dyspnoea severity [Modified Borg Scale (MBS)] and peripheral oxygen saturation were recorded. Pulmonary functions were assessed by spirometry.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years of age
* NYHA stage II-III
* LVEF of 45% or less
* Independently walking and climbing stairs
* Volunteer to participate in research

Exclusion Criteria:

* Any acute or chronic condition that would limit exercise capacity other than CHF
* Insufficient mental status to perform tests and surveys
* Orthopaedic problem limiting exercise test in lower extremity
* Severe obesity or there is a secondary cause for obesity
* Uncontrolled cardiac arrhythmia
* Unstable angina

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty-one patients age 65.52±7.57 years with stage II-III according to the NYHA classification, diagnosed with CHF, with a LVEF of 45% or less admitted to study.
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-12 (Actual)

PRIMARY OUTCOMES:
Symptom-Limited Stair-Climbing Test(SLSCT) | baseline
  predicted VO2 max (ml/kg/min)
Six-Minute Walk Test(6MWT) | baseline
  predicted VO2 max (ml/kg/min)
Cardiopulmonary Exercise Test(CPET) | baseline
  predicted VO2 max (ml/kg/min)

SECONDARY OUTCOMES:
Heart Rate | immediately after the procedure
  Heart Rate beats/min
Left Ventricular Ejection Fraction | baseline
  Ecocardiography
Blood Pressure | immediately after the procedure
  Systolic and diastolic blood pressure (mmHg)

OTHER OUTCOMES:
FVC l/sec | baseline
  Forced Vital Capacity l/sec
FEF 25-75 l/sec | baseline
  Forced Expiratory Flow 25-75 l/sec
PEF l/sec | baseline
  Peak Expiratory Flow l/sec
FEV1 % | baseline
  Forced Expiratory Volume in One Second %
FVC % | baseline
  Forced Vital Capacity %
FEF 25-75 % | baseline
  Forced Expiratory Flow %
PEF % | baseline
  Peak Expiratory Flow %
FEV1 l/sec | bseline
  Forced Vital Capacity l/sec
FEV1/FVC | bseline
  FEV1/FVC %